CLINICAL TRIAL: NCT00439660
Title: Double-Blind Randomized Placebo-Controlled Dose Escalating Phase Ib/IIa Study to Evaluate the Safety and Immunogenicity of Live Attenuated Oral Rotavirus Vaccine 116E in Healthy Non-Malnourished Infants 8 to 20 Weeks of Age
Brief Title: Dose Escalation Study to Evaluate Oral Rotavirus Vaccine 116E Live Attenuated in Healthy Infants 8 to 20 Weeks Old
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Collaborators: Ministry of Science and Technology, India (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); Stanford University (Other); Indian Council of Medical Research (Other Government); PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BBIL/ROTA/014; ISRCTN57452882 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Diarrhea
Keywords: Rotavirus, diarrhea, vaccine
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: Randomised double blind placebo controlled tri
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomised double blind placebo controlled tri

ARMS (2):
- rotavirus vaccine 116E 1 X 10(4) (Experimental): vaccine dose of 1 X 10(4) focus-forming units (ffu) in three doses starting at 6 weeks : 4 weeks apart each dose
  Interventions: Biological: Oral Rotavirus Vaccine 116E Live Attenuated
- rotavirus vaccine 116E 1 X 10(5) (Experimental): vaccine dose of 1 X 10(5) focus-forming units (ffu) in three doses starting at 6 weeks : 4 weeks apart each dose
  Interventions: Biological: Oral Rotavirus Vaccine 116E Live Attenuated

INTERVENTIONS:
Biological: Oral Rotavirus Vaccine 116E Live Attenuated

SUMMARY:
This study will be a Phase I, randomized, double blind, safety and immunogenicity trial of the Vero cell based 116E neonatal rotavirus vaccine candidate strain in healthy non-malnourished infants aged 8-20 weeks at three different dosage levels i.e.10^4.0, 10^5.0 and 10^6.0 FFU and for three administrations of each of these dosages given to infants at 4-week intervals. 180 infants (90 vaccinees/90 placebo) will be enrolled for each of the three dosage levels. The progression from the lower to the next higher dosage will be based on approval by the Data Safety Monitoring Board (DSMB) to be constituted by the Department of Biotechnology, New Delhi.

DETAILED DESCRIPTION:
Infants will be identified through a community survey in urban neighborhoods in the city of Delhi, India and screened at 6 weeks of age if parental consent is available. They will be given the first dose of EPI vaccines at this age. Of those screened, eligible infants will be given the first administration of the test vaccine/placebo at 8 weeks of age if they meet the enrollment inclusion criteria, and consent is available. The safety profile will be studied through daily home visits for 14 days post administration. Stool specimens will be collected before vaccination (day 0) and on days 3, 7 and 28 post administration of vaccine/placebo. Subsequently, two contacts will be made; a home visit on day 21 and a clinic visit on day 28. On the day 28 visit, a stool and blood specimen will be collected. Prior to each administration of vaccine/placebo the infants will be assessed for any contraindications.

All screened infants will be offered EPI vaccines as scheduled. The second and third administration of study vaccine/placebo will be at 12 and 16 weeks of age and the same strategy will be followed for each of the three dosages The study vaccine/placebo are not being administered with the EPI vaccines even though in the future rotavirus vaccine and the EPI vaccines may be coadministered. For the purpose of this study this schedule is being adopted, as no data are available on the interaction of EPI vaccines with this rotavirus vaccine candidate.

Baseline sera will be collected at 6 weeks (at the time of screening) and again 4 weeks after administration of the vaccine/placebo in a randomly selected subsample after the first (60 infants), second (60 infants) and third (60 infants) administration of each dosage.

Clinical adverse events will be monitored and relatedness to vaccine/placebo administration assessed for 14 days after each administration of the dosage under study, whereas monitoring for symptoms of intussusception will be assessed throughout the 28 day follow up period. Laboratory adverse events will be monitored for upto 28 days after first administration of each dosage. After the 4 week follow up of the third administration of the vaccine/placebo of the lowest dosage (10^4.0) is completed for all enrolled infants and the data safety monitoring board (DSMB) meeting will be convened and the data from the study will be analyzed, the code broken. If the DSMB declares the dosage safe, guided by the apriori criteria, the team will move on to screening infants for the next higher dosage (10^5.0) and the strategy listed above will be repeated for a total of 180 enrolled infants (90 vaccinees/90 placebo). The DSMB will again meet to review the data available from this cohort (i.e. 10^5.0) and the team will proceed to screen infants for the next higher dosage (10^6.0) only if the former is declared safe.

At the end of the study i.e. after the last visit of the last participant, based on reactogenicity and immunogenicity profile of each dosage, the appropriate dosage will be selected for further clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Access to telephone at home or in the immediate neighborhood.
2. Healthy male and female non-malnourished (weight for length not ≤ -3 SD of WHO child growth standards) infants aged 6 weeks (till 6 weeks + 2 days).
3. Parent's permission to participate in the study is available.
4. No plans to travel over the next 4 months

Exclusion Criteria:

1. Gestational age <37 weeks.
2. Any major physical congenital malformation.
3. Living in a household or has contact with an individual who is immunosuppressed.
4. Hospitalized once or more for the following illnesses since birth: heart disease, pneumonia, sepsis, meningitis, unconsciousness.
5. Is required to take daily medications other than vitamins or herbal "tonics".
6. Evidence of cardiovascular disease as indicated by any of the following:

   * Central cyanosis
   * Cyanotic or apnoeic spells
   * Features of congestive heart failure
   * Significant heart murmur detected on physical examination
7. Evidence of gastrointestinal disease indicated by following:

   * Diarrhea in the previous 7 days
   * Blood in the stools any time since birth
8. Evidence of neurological disease, as indicated by:

   * History of seizures any time since birth
   * History of unconsciousness
   * Focal deficit on physical examination
9. Evidence of liver or other reticuloendothelial disease, as indicated by any of the following:

   * Positive serology for hepatitis B surface antigen
   * Positive serology for hepatitis C antibody
   * SGOT or SGPT more than 1.25 times upper limit of normal (Upper limit normal SGOT 80 IU/L, SGPT 40 IU/L)
   * Alkaline phosphatase more than 1.25 times upper limit of normal (Upper limit of normal -470 IU/L)
   * Hepatomegaly (liver palpable 3 cm below costal margin), splenomegaly (palpable spleen), jaundice, or lymphadenopathy on physical examination
   * Serum bilirubin 1.25 times the upper limit of normal for age (Upper limit of normal 1.0 mg/dL).
10. Evidence of hematologic, rheumatologic, or immunologic disease, as indicated by any of the following:

    * Total leukocyte count <3500 or >15,000/mm3
    * Hemoglobin <9 g/dL or >17g/dL
    * Platelet count <100,000/mm3
    * Any episode of sepsis, pneumonia or meningitis requiring hospitalization since birth.
11. Evidence of renal disease as indicated by any of the following:

    * Creatinine >0.5 mg/dL
    * Hematuria (≥5 RBC/hpf)
    * Proteinuria (≥1+ per day)

Ages: 8 Weeks to 20 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
116E rotavirus vaccine | 6,10 and 14 weeks
  Safety

SECONDARY OUTCOMES:
116E rotavirus vaccine | 6,10 and 14 weeks
  immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Nita Bhandari, MBBS, PhD, Principal Investigator — Society for Applied Studies
Locations (1):
- Society for Applied Studies (SAS), New Delhi, India

REFERENCES:
- [Background] Bhandari N, Sharma P, Glass RI, Ray P, Greenberg H, Taneja S, Saksena M, Rao CD, Gentsch JR, Parashar U, Maldonado Y, Ward RL, Bhan MK. Safety and immunogenicity of two live attenuated human rotavirus vaccine candidates, 116E and I321, in infants: results of a randomised controlled trial. Vaccine. 2006 Jul 26;24(31-32):5817-23. doi: 10.1016/j.vaccine.2006.05.001. Epub 2006 May 12. PMID 16735085
- [Derived] Appaiahgari MB, Glass R, Singh S, Taneja S, Rongsen-Chandola T, Bhandari N, Mishra S, Vrati S. Transplacental rotavirus IgG interferes with immune response to live oral rotavirus vaccine ORV-116E in Indian infants. Vaccine. 2014 Feb 3;32(6):651-6. doi: 10.1016/j.vaccine.2013.12.017. Epub 2013 Dec 25. PMID 24374502
- [Derived] Bhandari N, Sharma P, Taneja S, Kumar T, Rongsen-Chandola T, Appaiahgari MB, Mishra A, Singh S, Vrati S; Rotavirus Vaccine Development Group. A dose-escalation safety and immunogenicity study of live attenuated oral rotavirus vaccine 116E in infants: a randomized, double-blind, placebo-controlled trial. J Infect Dis. 2009 Aug 1;200(3):421-9. doi: 10.1086/600104. PMID 19545211